CLINICAL TRIAL: NCT06967285
Title: Changes in Cerebral Blood Flow Before and After Prone Position in Patients With ARDS Predict the Occurrence of Neurological Complications
Brief Title: Prone Positioning in ARDS: Predicting Neurological Complications Via Cerebral Hemodynamics
Acronym: PRONEBRAINAR
Status: Recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Lingai Pan, Deputy Chief Physician, Sichuan Provincial People's Hospital
Other Study IDs: KY2025PD21
Record Dates: First submitted 2025-03-22; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: ARDS (Moderate or Severe)
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Prone ventilation — Cerebral Blood Flow Monitoring Before and After Prone Ventilation in Patients with ARDS.Cerebral blood flow,intracranial pressure,and systemic hemodynamic monitoring were performed at the following time points:before prone positioning(T0),1 hour after prone ventilation(T1),12 hours after prone ventilation(T2),1 hour after returning to the supine position(T3),and 7 days after returning to the supine position(T4).

SUMMARY:
Prone Positioning in ARDS: Predicting Neurological Complications via Cerebral Hemodynamics

DETAILED DESCRIPTION:
Collecting Medical Records, Demographic Characteristics, and Clinical Data of Moderate to Severe ARDS Patients Requiring Prone Positioning Treatment at Chengdu Pixdu District People's Hospital, Sichuan Provincial People's Hospital, The Fourth People's Hospital of Chengdu, and Chengdu Shuangliu District First People's Hospital from March 2025 to March 2026.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* Meet the diagnostic criteria for ARDS(Acute Respiratory Distress Syndrome),with PaO₂/FiO₂<150 mmHg,and requiring prone ventilation
* Expected duration of mechanical ventilation>48 hours
* Written informed consent obtained

Exclusion Criteria:

* Presence of contraindications to prone positioning(e.g.,head and neck injuries,spinal instability,severe intracranial hypertension)
* Severe neurological diseases(e.g.,cerebral hemorrhage,cerebral infarction,intracranial space-occupying lesions)that may affect the monitoring of cerebral hemodynamics
* Life-threatening ARDS
* Patients who are unable to undergo neurological assessment
* Poor image quality or absence of images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Moderate to Severe ARDS Expected to Undergo Mechanical Ventilation for Over 48 Hours
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Neuroimaging Studies | From enrollment to 2 weeks after the end of treatment.
  Cranial CT or MRI Scans Conducted Before and After Prone Positioning to Detect New-Onset Neurological Complications Such as Cerebral Edema, Intracranial Hemorrhage, and Cerebral Infarction
Biomarker Detection | From enrollment to 2 weeks after the end of treatment.
  Blood samples were collected for NSE(Neuron-specific Enolase)and IL-6(Interleukin-6)before and after prone positioning.

SECONDARY OUTCOMES:
Incidence rate of delirium | From enrollment to 2 weeks after the end of treatment.
  Assessment using the Confusion Assessment Method for the Intensive Care Unit(CAM-ICU)was conducted before and after prone position therapy in patients.
Cognitive function | From enrollment to 2 weeks after the end of treatment.
  Assessment using the Mini-Mental State Examination(MMSE)was conducted before and after prone position therapy in patients.

CONTACTS AND LOCATIONS:
Overall Officials: lingai Pan, PhD, Study Chair — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital,, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No